CLINICAL TRIAL: NCT00001046
Title: Active Immunization of HIV-Infected Pregnant Women: A Phase I Study of Safety and Immunogenicity of a rgp120/HIV-1 Vaccine (NOTE: Some Patients Receive Placebo)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Prevention
Other Study IDs: ACTG 233; 11210 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy; HIV Seronegativity
Keywords: Vaccines, Synthetic; Pregnancy; Pregnancy Complications, Infectious; AIDS-Related Complex; HIV Envelope Protein gp120; HIV Preventive Vaccine; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious; AIDS-Related Complex | interventions — MF59 oil emulsion

INTERVENTIONS:
Biological: MF59
Biological: rgp120/HIV-1 SF-2

SUMMARY:
PRIMARY: To evaluate the short-term safety of rgp120/HIV-1SF2 vaccine versus MF59 placebo administered to HIV-infected pregnant women.

SECONDARY: To evaluate the immunogenicity and long-term safety of rgp120/HIV-1SF2 in HIV-infected pregnant women who received the vaccine during pregnancy only or during pregnancy and postpartum. To evaluate immunogenicity and safety in the infant through 18 months of age following maternal immunization with the vaccine during pregnancy.

Active immunization of HIV-infected women during pregnancy may slow the progression of maternal disease, reduce the titer of virus in maternal plasma, and increase the titer of epitope-specific antibody. Also, active immunization has the potential to induce primary immunity in the fetus and to boost both T-cell and humoral immune responses to HIV in the mothers.

DETAILED DESCRIPTION:
Active immunization of HIV-infected women during pregnancy may slow the progression of maternal disease, reduce the titer of virus in maternal plasma, and increase the titer of epitope-specific antibody. Also, active immunization has the potential to induce primary immunity in the fetus and to boost both T-cell and humoral immune responses to HIV in the mothers.

Women are randomized to receive rgp120/HIV-1SF2 vaccine or MF59 placebo. Patients receive the first immunization between 16 and 24 weeks gestation and monthly thereafter until delivery, for a maximum of five immunizations. Patients may continue to receive the immunization regimen to which they were originally assigned at 3, 6, 9, and 12 months postpartum. Maternal follow-up continues until 18 months postpartum; infants are followed until age 18 months.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed during pregnancy:

* AZT.
* Methadone maintenance.

NOTE:

* Patients may not initiate antiretroviral therapy for disease progression.

NOTE:

* Patients may change from AZT to another antiretroviral agent or may begin antiretroviral therapy following delivery, if clinically indicated.

Patients must have:

* Documented HIV infection.
* CD4 count >= 400 cells/mm3 (average of two determinations obtained 1 week apart).
* No clinical criteria for a diagnosis of AIDS.
* HIV p24 antigen <= 30 pg/ml.
* Estimated gestational age between 16 and 24 weeks, confirmed by baseline sonogram that does not demonstrate any congenital abnormalities considered to be incompatible with life.
* Intention to carry pregnancy to term.
* Willingness to be followed by an ACTU for the duration of the study.

NOTE:

* Father of the fetus (if available after a reasonable attempt to contact him) must provide informed consent.

Prior Medication:

Allowed:

* AZT.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known hypersensitivity to a component of the vaccine.
* Hepatitis B antigen positive at study entry.
* Evidence of life-threatening or other serious pre-existing fetal abnormalities (e.g., anencephaly, renal agenesis, Potter's syndrome).
* Evidence of syphilis that requires therapy during this pregnancy.
* Intention to breast-feed.

Presence of obstetrical high-risk factors such as:

* insulin-dependent diabetes
* hypertension requiring the use of anti-hypertensive therapy
* repeated intrauterine fetal demise
* Rh-sensitization or other blood group alloimmunization
* diseases requiring use of immunosuppressive therapy (e.g., asthma, lupus).

Concurrent Medication:

Excluded during pregnancy:

* Antiretrovirals other than AZT.
* Immunomodulating agents (e.g., HIVIG, IVIG).
* Other investigational drugs or immunosuppressive agents.

NOTE:

* Patients may change from AZT to another antiretroviral agent or may begin antiretroviral therapy following delivery, if clinically indicated.

Prior Medication:

Excluded within 90 days prior to study entry:

* Antiretrovirals other than AZT.
* Immunomodulating agents (e.g., HIVIG, IVIG).

Current use of illicit drugs or chronic alcohol use by patient history.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Starr S, Study Chair; Allen M, Study Chair; Scott GB, Study Chair; Silverman N, Study Chair